CLINICAL TRIAL: NCT06508827
Title: Iron With Standard of Care Immunotherapy in Melanoma
Brief Title: Intravenous Iron in Combination With Standard of Care Immunotherapy in Melanoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty recruiting participants
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Mateusz Opyrchal, Associate Professor of Medicine, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTO-IUSCCC-0854
Record Dates: First submitted 2024-07-15; First posted 2024-07-18 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Anemia, Iron Deficiency; Melanoma
Keywords: Erythroid Progenitor Cells; Iron; Anemia; Melanoma
MeSH Terms: conditions — Anemia, Iron-Deficiency; Melanoma; Anemia | interventions — Iron-Dextran Complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Iron dextran 1000 mg IV (Experimental): Iron dextran 1000 mg IV will be administered once, about 7 days prior to standard of care treatment.
  Interventions: Drug: Iron dextran 1000 mg IV

INTERVENTIONS:
Drug: Iron dextran 1000 mg IV — Iron dextran 1000 mg IV will be administered once, about 7 days prior to standard of care treatment.

SUMMARY:
Anemia is a common complication among cancer patients and is negatively associated with overall prognosis and therapeutic outcomes. The purpose of this study is to see if giving a dose of iron prior to any standard of care chemotherapy treatment will affect the cells that are believed to make treating melanoma harder, making melanoma more responsive to the standard of care immunotherapy.

DETAILED DESCRIPTION:
This is a pilot single arm, non-randomized study involving adult patients with melanoma receiving standard of care treatment with hemoglobin levels less than 13 g/dl, ferritin levels below 100 ng/ml, and transferrin saturations of less than 30%.

Cancer-associated anemia remains an underestimated and inadequately treated chronic condition that adversely affects the quality of life and overall prognosis in cancer patients. The correction of anemia in cancer patients would be a clinically applicable strategy to prevent and/or mitigate the expansion of tumor promoting erythroid progenitor cells (EPCs). Iron is an essential functional component of erythrocyte hemoglobin and is a crucial regulator of erythropoiesis. Strategies to therapeutically target the immunosuppressive machinery have emerged as a promising approach for cancer treatment. By promoting EPCs differentiation/maturation in anemic melanoma patients, immunosuppression could be mitigated and the therapeutic activity of immune checkpoint inhibitors enhanced.

A dose of intravenous iron will be given one week prior to standard of care chemotherapy and antibodies CD71 and CD235a will be used to detect EPCs in circulation and tumor microenvironment.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old adults at the time of informed consent
2. Ability to provide written informed consent and HIPAA authorization
3. Biopsy confirmed melanoma
4. Eligible for standard of care treatment
5. Plan to undergo immunotherapy in neoadjuvant or metastatic setting
6. ECOG performance status 0-2
7. Anemia defined as hemoglobin < 13 g/dl in addition to ferritin < 100 ng/ml and/or transferrin saturation < 30%

Exclusion Criteria:

1. History of anaphylactic reaction to intravenous iron or any proposed standard of care treatments
2. Diagnosis of hemoglobinopathies
3. Therapeutic Iron supplementation in the past 3 months (oral iron as part of MVI allowed)
4. Diagnosis of hemochromatosis
5. Symptomatic brain metastases that require local treatment (brain metastasis which will be treated with systemic immunotherapy or treated metastasis with without need for steroids for symptomatic management are eligible).
6. Pregnant or lactating female adults
7. Active infections which in research teams' opinion increases risk for toxicities
8. Any condition that in the opinion of PI may interfere with patient being able to complete the required procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Erythroid progenitor cells (EPCs) detection in patient's blood | Baseline, 1 week post iron infusion, 21 days post iron infusion
  Whether the erythroid progenitor cells (EPCs) can be detected at baseline in patient's blood in 3 out of 5 evaluable patients

SECONDARY OUTCOMES:
Iron dose tolerance | baseline
  At least 50% of patients consented successfully receive >50% of planned iron infusion

CONTACTS AND LOCATIONS:
Overall Officials: Mateusz Oprychal, MD, PhD, Principal Investigator — Indiana University

IPD SHARING:
Plan to Share IPD: Undecided